CLINICAL TRIAL: NCT05327127
Title: Study to Evaluate the Efficacy and Safety of Combination Therapy of K-877-ER and CSG452 in Participants With Noncirrhotic Nonalcoholic Steatohepatitis (NASH) With Liver Fibrosis
Brief Title: Study to Evaluate the Efficacy and Safety of K-877-ER and CSG452 in Participants With NASH With Liver Fibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-001-201
Record Dates: First submitted 2022-03-02; First posted 2022-04-14 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: NASH
MeSH Terms: interventions — 6-((4-ethylphenyl)methyl)-3',4',5',6'-tetrahydro-6'-(hydroxymethyl)spiro(isobenzofuran-1(3H),2'-(2H)pyran)-3',4',5'-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- K-001 (Experimental): K-877-ER and CSG452 Once daily (QD)
  Interventions: Drug: K-877-ER; Drug: CSG452
- K-877-ER (Experimental): K-877-ER and CSG452 Placebo QD
  Interventions: Drug: K-877-ER; Drug: Placebo
- CSG452 (Experimental): CSG452 and K-877-ER Placebo QD
  Interventions: Drug: CSG452; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K-877-ER — K-877-ER tablet
  Arms: K-001; K-877-ER
Drug: CSG452 — CSG452 tablet
  Arms: CSG452; K-001
Drug: Placebo — Placebo tablet
  Arms: CSG452; K-877-ER; Placebo

SUMMARY:
A study to investigate the use of combination therapy with two investigational products for the treatment of adult patients with Nonalcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with study procedures and give written informed consent
* Age ≥18 years
* NAS ≥4 with a score of at least 1 in each component of the NAS (steatosis, lobular inflammation, and ballooning) at Visit 2 liver biopsy, or a historical liver biopsy performed within 24 weeks of randomization
* Fibrosis stage of 1 or greater and below 4 on NASH CRN (Clinical Research Network) fibrosis staging system at Visit 2 liver biopsy, or a historical liver biopsy performed within 24 weeks of randomization
* Meet all inclusion criteria outlined in clinical study protocol

Exclusion Criteria:

* Participation in another clinical trial involving an investigational agent within 30 days prior to signing the Informed Consent Form (ICF) for this study
* Ongoing or recent consumption of Greater than moderate amounts of alcohol as defined in clinical study protocol
* Evidence of other forms of chronic liver disease as defined in clinical study protocol
* Does not meet any other exclusion criteria outlined in clinical study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in disease activity and no worsening of liver fibrosis (Yes/No) | Baseline to Week 48
  The improvement in disease activity is defined as decrease in NAFLD Activity Score (NAS) ≥2 points. The worsening of fibrosis is defined as any numerical increase in the stage.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events (AE) | 52 Weeks
  Time frame is 52 weeks unless an unresolved AE is still being followed

CONTACTS AND LOCATIONS:
Overall Officials: Shona Pendse, MD, MMSc, Study Chair — Kowa Research Institute, Inc.
Locations (77):
- United States (37):
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Arcare Center for Clinical Research, Little Rock, Arkansas
  - Clinical Trials Research, Lincoln, California
  - United Clinical Research Institute, Los Alamitos, California
  - Velocity Clinical Research, Los Angeles, California
  - Alliance Clinical Research, Poway, California
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - ENCORE Borland Groover Clinical Research, Jacksonville, Florida
  - Miami Clinical Research, Miami, Florida
  - Ocala GI Research, Ocala, Florida
  - Sensible Healthcare Clinical Research, LLC, Ocoee, Florida
  - Centricity Research, Columbus, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Iowa Digestive Disease Center, Clive, Iowa
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Mid-Atlantic GI Research, LLC, Greenbelt, Maryland
  - Boston Medical Center Boston University Chobanian & Avedisian School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - GI Alliance Research, Flowood, Mississippi
  - GI Associates Research, LLC, Columbia, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Lucas Research, Inc., Morehead City, North Carolina
  - DSI Research Northridge, LLC, Dayton, Ohio
  - Penn State Health/Penn State College of Medicine, Hershey, Pennsylvania
  - GI Alliance Research, Cedar Park, Texas
  - GI Alliance Research, Dallas, Texas
  - GI Alliance Research, Garland, Texas
  - GLRI McAllen Research, Pharr, Texas
  - Northeast Clinical Rsearch of San Antonio, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Impact Research Institute, Waco, Texas
  - Digestive Health Research of Central Texas, LLC, Waco, Texas
  - North Richmond Health Research, Richmond, Virginia
  - GI Select Health Research, Richmond, Virginia
  - Centricity, Suffolk, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Argentina (6):
  - Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - CINME - Centro De Investigaciones Metabolicas, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas de Mar del Plata, Mar del Plata, Buenos Aires
  - Hospital Universitario Austra, Pilar, Buenos Aires
  - Hospital Provincial del Centenario, Santa Fe, Rosario
- Brazil (4):
  - Clínica de Endocrinologia e Metabologia Ltda, Brasília, Brasilia DF
  - Hospital Alianca Rede D 'Or, Salvador, Estado de Bahia
  - Hospital Universitário João de Barros Barreto, Belém, Pará
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Porto Alegre RS
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Ecogene-21, Chicoutimi, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Japan (23):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Ehime University Hospital, Tōon, Ehime
  - Fukui-ken Saiseikai Hospital, Fukui-shi, Fukui
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - NHO Takasaki General Medical Center, Takasaki Shi, Gumna
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima, Hiroshima
  - NHO Kure Medical Center and Chugoku Cancer Center, Kure Shi, Hiroshima
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - JCHO Hokkaido Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - SHIN-YURIGAOKA General Hospital, Kawasaki, Kanagawa
  - St. Marianna University School of Medicine, Kawasaki, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Tohoku Rosai Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto Shi, Nagano
  - Nagano municipal Hospital, Nagano, Nagano
  - Saiseikai Niigata Hospital, Niigata, Niigata
  - Kawasaki Medical School General Medical Center, Okayama, Okayama-ken
  - Saga University Hospital, Saga, Saga-ken
  - Japanese Red Cross Musashino Hospital, Musashino, Tokyo
  - Nippon Medical School Hospital, Bunkyō City, Toyko
  - Oita Cardiovascular Hospital, Ōita
- Spain (4):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Puerta De Hierro, Madrid